CLINICAL TRIAL: NCT03022058
Title: Evaluation of the EarEEG System for Detection of Hypoglycaemia-induced Changes in the EEG in Subjects With Type 1 Diabetes: A Non-controlled, Exploratory Study
Brief Title: Evaluation of the EarEEG System for Detection of Hypoglycaemia-induced Changes in the EEG in Subjects With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Aarhus (Other); T&W Engineering A/S (Industry); UNEEG Medical A/S (Industry)
Responsible Party: Principal Investigator, Henning Beck-Nielsen, Professor, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 56205
Record Dates: First submitted 2016-12-13; First posted 2017-01-16 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with type 1 diabetes mellitus (Experimental)
  Interventions: Device: Ear-EEG system

INTERVENTIONS:
Device: Ear-EEG system — Measurement of the neural activity in the brain by use of the Ear-EEG device, which is a customized earplug containing 6 embedded dry electrodes placed inside the ear canal and in the concha of the ear.

SUMMARY:
The EarEEG system is a novel non-invasive, unobstructed and discrete method for recording EEG in which the signal is recorded using dry-contact electrodes embedded on a customised ear piece. One intended medical indication of the EarEEG system is the detection of hypoglycaemia-induced changes in the EEG in patients with type 1 diabetes. Currently, no studies exist investigating the detection of hypoglycaemic episodes by use of ear electrodes. While a finger prick test accurately measures the blood glucose level, it does not provide continuous measurements, and hence it is unreliable as a hypoglycaemia alarm. Recent studies have indicated that the use of continuous glucose monitoring (CGM) reduces the risk of severe hypoglycaemia. However, some find these devices troublesome to use and utilisation of CGM has remained limited to date. Observational data show that only a small percentage of patients with type 1 diabetes are using CGM on an ongoing basis. Thus, there is a medical need for a reliable hypoglycaemia detection device which is easy and convenient to use.

This clinical study aims at investigating the feasibility of measuring hypoglycaemia induced changes in the EEG by use of the EarEEG system.

ELIGIBILITY:
Inclusion Criteria:

For a subject to be eligible, all inclusion criteria must be answered "yes":

1. Informed consent obtained before any study related activities1
2. Age 18-70 years
3. Patients with type 1 diabetes (duration ≥ 5 years)

Exclusion Criteria:

For a subject to be eligible, all exclusion criteria must be answered "no":

1. Severe cardiac disease

   1. History of myocardial infarction
   2. Cardiac arrhythmia
2. Previous stroke or cerebral haemorrhage and any other structural cerebral disease
3. Uraemia defined as s-creatinine ≥ 3 times upper reference value,
4. Liver disease defined as s-ALAT ≥ 3 times upper reference interval
5. Epilepsy
6. Use of antiepileptic drugs for any purposes
7. Use of the following drugs: Chemotherapeutic drugs of any kind, methotrexate, third generation antipsychotic drugs (aripiprazole, quetiapine, clozapine, ziprasidone, paliperidone, risperidone, sertindole, amisulpride, olanzapine)
8. Known or suspected abuse of alcohol defined as estimated consumption beyond that, which is recommended by the DHA1 or any other neuro-active substances
9. Use of hearing aid or cochlear implants2
10. Allergic contact dermatitis caused by metals or generally prone to skin irritation
11. Narrow or malformed ear canals
12. Patients that are judged incapable of understanding the patient information or who are not capable of carrying through the investigation
13. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Presence of significant qEEG hypoglycaemia indicators when comparing normo- and hypoglycaemic EEG as measured by the EarEEG systems for subjects where hypoglycaemia-induced changes have been observed in the scalp EEG (visit 4) | Up to 8 hours
  During insulin-induced hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Henning Beck-Nielsen, DMSc, Principal Investigator — Odense University Hospital
Locations (1):
- Diabetes Research Center, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided